CLINICAL TRIAL: NCT06343675
Title: Systematic Health-promoting Work Environment Management in Dentistry - Workplace Interventions and Work Adjustments for Dental Health Professionals
Brief Title: Systematic Health-promoting Work Environment Management in Dentistry
Status: Completed | Type: Observational
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Anneli Peolsson, Professor, PhD, MSc PT, MSc HRMD, Linkoeping University
Other Study IDs: Dnr 2024-00620-01
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Occupational Health
Keywords: Dental staff, workplace

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cross-sectional study with sub-group interviews: Dental staff
  Interventions: Other: There is no intervention

INTERVENTIONS:
Other: There is no intervention — There is no intervention

SUMMARY:
Research shows that the workplace is an important arena where much can be done to promote a sustainable working life while maintaining health. However, there is a lack of knowledge that is specific to dental care with regard to managers' and employees' perceptions of the work environment, systematic work environment management and work adaptations, as well as what measures in the workplace are necessary to create a health-promoting and sustainable work environment. There is also a lack of knowledge regarding what support employees and managers need in the systematic work environment management and what individual workplace adaptations that can work within dental care organizations.

DETAILED DESCRIPTION:
There is a lack of information about how systematic work environment management works in dental care. This includes the dental staff's and management's experience of how and how well systematic health-promoting work environment management is applied, what individual workplace adaptations are used, what support they lack and what they think is good regarding the work environment management. The dental work environment includes dentists, dental hygienists and dental nurses. Perceptions of the work environment and work-related interventions are poorly studied.

Overall aim: Based on a health-promoting basis, the research project aims to study conditions in the work environment in dental care and what support is needed in the systematic work environment management.

Sub-study one is a quantitative cross-sectional study and sub-study two is a qualitative interview study.

Sub-study 1

Aim, sub-study 1: The aim is to investigate how employees and managers in dental care perceive their work environment, support in the organization, safety at work and the need for work environment measures and work adaptations. Furthermore, the aim is to map the employees' self-rated health. The study also aims to describe how managers perceive opportunities to actively work with systematic work environment management in dental care.

Research questions in sub-study 1:

* How do dental staff estimate perceived physical and mental health and work ability?
* Are there differences between those who have good health, musculoskeletal illness and mental illness with regard to perceptions of the work environment? How is the need for support for systematic work environment management described, including individual workplace adaptations among employees and managers?

Participants: Employees and managers in dental care. The goal is to recruit at least 200 dental professionals.

Inclusion criteria are to have employment (or self-employed) as a dentist, dental hygienist, dental nurse, clinic coordinator or operations manager in private or public dental care. All employees are included, including those on sick leave and parental leave, regardless of their level of work and employment. There is no exclusion criteria, those working in dental care had to understand the Swedish language and will thereby be able to understand the survey/questions.

Recruitment: The study is national and recruitment takes place in all regions in Sweden with a selective selection where the goal is to get a wide range of respondents in different counties. Brief information about the project and a QR code for the project's website will be disseminated through advertising in various media channels, intra-regional mailings, digital platforms and personal contacts. The investigators will also disseminate information to prospective participants via the trade unions, HR and managers. In addition, contact persons at various dental clinics and trade unions will assist with the distribution. On the website, detailed information about the study is available to give prospective participants an understanding of the purpose of the study and how their data will be processed. Participants are informed to give their consent to participate in the study by answering the first question in the survey.

The data collection consists of a digital survey in the digital tool Webropol, which is answered via an open link on the project's website.

The questionnaire contains questionnaires that measure perceived work ability, health, work-related problems, pain, stress, sleep, productivity and a questionnaire for the study. Background questions such as occupation, type of employment, age, family situation and issues related to perceptions of safety at work, the need for work environment measures and workplace adaptations, as well as opportunities to receive and provide support in this area, are also included. Open-ended questions are asked about their experience of work environment management at the workplace and what support they would like to see. Before the cross-sectional study is conducted, the questionnaire is tested in a smaller pilot study to ensure that it is not too long or difficult to answer. For managers, the survey also contains questions about the conditions for taking responsibility for and driving systematic work environment management and individual work adaptations, as well as what support they would like. The questionnaire ends with a question about whether they are interested in participating in sub-study 2 (link to participant information is available and contact information for the project member) and in any contact for a follow-up study. If participants are interested in this, they are asked to provide their name, social security number and contact details. Those who do not want to provide personal data are anonymous (i.e. the researchers do not know their name and contact details, theoretically the IP address could be traced but we do not intend to do so / knowledge and therefore consider the participants anonymous).

Analysis: Data will be analyzed using descriptive statistics (mean and spread), correlation analyses where independent t-test and Mann-Whitney U-test will be used. Correlation and regression analyses are also used in the analyses. Furthermore, the responses from different subgroups of employees (gender, type of work, degree of anxiety/depression) will be analyzed to understand possible variations regarding the relationship between work ability, work-related problems and the systematic work environment management.

The hypothesis is that with a lower assessment of work ability, higher demands at work and a higher estimation of work-related problems, the greater the importance of the opportunities for work adaptations at work and a well-executed systematic work environment management.

For this study, power is based on work ability single item, with a 90% power and effect size of 0.5. A difference in average with three steps and spread of 1, we need at least 70 employees and managers/clinic coordinators. To enable subgroup analyses, at least 200 people will be recruited.

Open-ended questions are analyzed with content analysis.

Sub-study 2

Purpose of sub-study 2: The aim is to explore managers' perceptions of systematic work environment management, their role in and experiences of systematic work environment management and what need for support participants have to be able to work with health promotion.

Research questions in sub-study 2:

* How do managers in dental care experience a health-promoting and good work environment?
* What in the business do the managers perceive to be the greatest risks of ill health?
* What experiences do they describe of systematic work environment management?
* What support would they like in the systematic work environment management?

Recruitment: Managers from sub-study 1. Managers are recruited through a strategic selection principle in order to obtain as broad a description of perceptions as possible. Possible factors such as gender, age, professional experience, size of the business may be relevant for the selection. The investigators also want to include both private and public activities in different regions. Information about the project will be disseminated through contact persons in dental care and digitally. Contact persons ask prospective participants about their interest in participating and to provide contact information for the research group. Information will also be disseminated via digital channels such as social media (X, Facebook, LinkedIn) (appendix 2) and via blogs. People who are interested in participating can read more about the project and register their interest by filling out a digital form on the project's website. Thereafter, after the expression of interest, the research group contacts interested persons to provide further information about the study and obtain informed consent.

Data collection: Individual semi-structured interviews (see appendix 3) with managers and clinic coordinators in dental care will be conducted digitally through audio recording only. An interview guide on the areas to be covered (see Annex 3) will be tested in 2-3 pilot interviews. Background questions and open questions.

Interview guide:

Background data: age, gender, profession, year within the profession, year as a manager

1. Can you describe your role and mission? (On a general level)
2. Can you describe your role and mission with regard to the work environment?
3. How do you see the relationship between health and work environment?
4. What do you think a satisfactory and healthy work environment can look like in your business?
5. Can you describe your experiences of systematic work environment management (SAM) in your organisation?

   * Can you give some examples where it worked well?
   * Which interventions do you think have helped (the most)?
   * How do you see the work on the application of SAM in your business? (Challenges)
   * How do you feel about being able to support your employees in continuing and functioning at work or returning to work? (Linked to possible challenges and need for support?)
6. A. Can you describe your experiences of providing support in rehabilitation and individual workplace adaptations? B. Can you describe how you feel that the employees' need for work adaptation looks like in your business?

   * Can you give some examples where it worked well?
   * Which interventions do you think have helped (the most)?
   * Can you describe situations when it felt difficult or didn't turn out as planned? (Challenges, obstacles).
   * Based on your role of responsibility, how do you see any need for support for systematic work environment management and health-promoting work environment for all employees? (Linked to any challenges, employees' need for support, your need for support)
7. Is there anything else that you would like to bring up regarding your role in and experiences of systematic work environment management that we have not discussed?

Analysis: The interviews are transcribed verbatim and analyzed with content analysis.

ELIGIBILITY:
Inclusion Criteria:

* To have employment (or self-employed) as a dentist, dental hygienist, dental nurse, clinic coordinator or operations manager in private or public dental care.
* All employees are included, including those on sick leave and parental leave, regardless of their level of work and employment.

Exclusion Criteria:

* None. (To be able to work in a dental health care profession in Sweden it is a requirement to understand the Swedish language, language will therefore not be a criteria).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Employment (or self-employed) as a dentist, dental hygienist, dental nurse, clinic coordinator or operations manager in private or public dental care
Sampling Method: Non-Probability Sample
Enrollment: 732 (Actual)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Work Ability Single Item Scale (WAS) | descriptive data at baseline= one measurement
  Current workability compared with lifetime best WAS (score 0-10). and physical and mental demands in work
Work Ability physical demands | descriptive data at baseline= one measurement
  How do you assess your current work ability in relation to the physical demands of your job? Very good(5); Quite good (4) Moderate (3) Quite bad (2), Very bad (1)
Work Ability mental demands | descriptive data at baseline= one measurement
  How do you assess your current work ability in relation to the mental demands of your job? Very good(5); Quite good (4) Moderate (3) Quite bad (2), Very bad (1)
Sick leave | descriptive data at baseline= one measurement
  How many days have you been absent from work due to illness or injury related to work-related ill health in the past year (12 months)? No days; 1-7 days; 8-24 days; 25-99 days; 100-365 days

SECONDARY OUTCOMES:
Structured Multidisciplinary Work Evaluation Tool (SMET) | descriptive data at baseline= one measurement
  Structured multidisciplinary work evaluation tool, (SMET) will be used. The questionnaire asks about physically, environmentally and psychosocially demanding work items (30 items). A scale of 1-10 is used in the questionnaire, 1 is labeled "Not at all" and 10 is labeled "Highly".
Satisfaction with work | descriptive data at baseline= one measurement
  How satisfied are you with your work (0-5)
Global Health | descriptive data at baseline= one measurement
  General self-reported health obtained by the question: "In general, would you say your health is…?", with five anchor points ranging between excellent and poor
Perceived stress | descriptive data at baseline= one measurement
  Perceived stress obtained by the question: Stress refers to a situation where one feels tense, restless, nervous, or worried, or cannot sleep at night because they are constantly thinking about problems. Have you felt stressed recently? with five anchor points ranging between not at al (1) to very much (5)
Health problems related to work | descriptive data at baseline= one measurement
  Do you experience any discomfort related to work and tasks in your current profession? (You can provide multiple options); Face, jaws, Neck, Shoulder/Shoulders, Elbow/Elbows, Wrists/Hands, Thoracic spine, Lumbar spine, Hips, Knees, Ankles/Feet, Headache, Stress-related issues, Sleep difficulties, Anxiety, Exhaustion, Depression, Other, namely
Pain during last 7 days | descriptive data at baseline= one measurement
  Have you experienced any discomfort (pain, ache, discomfort) from your body at any time during the past 7 days? Yes/no. If Yes, scale, 0 = No discomfort and 10 Symptoms as severe as they can ever be
Psychological safety | descriptive data at baseline= one measurement
  Do you feel secure enough in the work group to dare to say what you think, question, or have a different opinion than the group? scale from "Not at al secure" (1) to "Completely secure" (10)
Work environment problems | descriptive data at baseline= one measurement
  Have you experienced any issues in your work environment in the past seven days? By work environment issues, we mean any potential physical, psychological, or social problems that may arise in the workplace. No/Yes In the past seven days, to what extent did work environment-related issues affect your work performance? Please check the appropriate number.
  0 means work environment issues did not affect my work performance 10 means work environment issues completely hindered me from working
Health related problems | descriptive data at baseline= one measurement
  Have you experienced health issues in the past seven days but still chose to go to work? By health issues, we mean any physical or emotional problems or symptoms. No/yes In the past seven days, to what extent did health issues affect your work performance? Please check the appropriate number.
  0 means health issues did not affect my work performance. 10 means health issues completely hindered me from working.
  Open question: If you have indicated health issues, what personal strategies do you have to be able to work despite these issues? Please describe them
Questions about workplace improvements, work adjustments, and support in the workplace | descriptive data at baseline= one measurement
  Open questions Do you have any suggestions on how your work environment can be improved at your workplace? If yes, describe how.
  If you have received work adjustments in your job, describe 1) what they were and 2) if they have been helpful to you.
Work adjustment and discomfort | descriptive data at baseline= one measurement
  In what ways do you have the opportunity to adjust your work on days when you feel discomfort? Scale: Always, sometimes, never
  Items:
  Can perform necessary work and postpone the rest Can choose among tasks Can receive help from colleagues Can work at a slower pace than usual Can take longer breaks Can shorten the workday Can use tools or equipment
  Open question: Are there other opportunities to adjust your work within dentistry? If yes, describe what they are.
  Open question: What support and work adjustments would you like from your immediate supervisor? If yes, describe what and how.
Support and meaning in work | descriptive data at baseline= one measurement
  Experience of support and meaning in work. Take a position on the following statement Scale: 1 - Strongly disagree; 2 - Disagree; 3 - Agree; 4 - Strongly agree
  Statements:
  My immediate supervisor cares about my health and well-being. Special efforts are made at my workplace to adapt working conditions based on employees' age.
  I feel sufficient support from my coworkers in my work. The social participation present at my workplace makes me want to stay. In my profession, it is desirable for older employees to stay as long as possible.
  I experience joy in my daily work. Work is important in my life. I have sufficient opportunities to participate in skills development. I find my work stimulating.
Sustainable work life | descriptive data at baseline= one measurement
  Sustainable work life. What do you think increases the possibility of being able to work until 69 years or longer. Take a position on the following statement; Opportunity for customized tasks based on my abilities, Workplace wellness activities, Reduction of physical job demands, Increased variation/rotation work tasks, Do Different tasks at work, Reduction job demands, Increased autonomy, More recovery time, Reduced work pace, Changes to the scheduling of working hours, Shorter work hours, Higher salary, accommodate different needs at different ages, Increased involvement in decision-making and organization of work, Opportunity for new knowledge/skill, New job within my profession and different profession
  Scale: 1 - Strongly disagree; 2 - Disagree; 3 - Agree; 4 - Strongly agree
Systematic work environment management and safety | descriptive data at baseline= one measurement
  How do you perceive that the employees at your workplace work according to systematic work environment management? 12 statements: Scale "Does not apply at all" to "Fully applies" the statetement concerns following areas: Prevention of injuries, Systematic work environment management, Procedures for conducting risk assessments, Use action plan, Safety behaviour and learn from experiences to prevent accidents, Safety representative role in prevention, Regular training to learn about work environment specifically tailored to dentistry.
Targeted questions to managers | descriptive data at baseline= one measurement
  F1. Do you have managerial responsibilities? No/Yes If yes, we ask you to answer the following questions related to your managerial responsibilities.
  F2. Questions for you as a manager about work environment responsibility Do you have work environment responsibility in your organization? Yes/No
  Is the work environment responsibility clearly delegated?Yes,To some extent. No
Work environment responsibility and measures | descriptive data at baseline= one measurement
  Do you feel that as a manager, you have sufficient knowledge to take on work environment responsibility? Do you have resources to implement measures? Do you have the authority to decide on measures? Do you have the opportunity to be present as a manager and lead the work for a good work environment?
  Scale: Not at all (1)Very much (10)
Work environment management support and education | descriptive data at baseline= one measurement
  Open questions:
  Do you, as a manager, need training to take responsibility for systematic work environment management and work adjustments? If yes, what type of training do you need?
  Do you, as a manager, need support in systematic work environment management? If yes, describe what type of support.
  Is there anything else you would like to convey as a manager regarding the conditions for a good work environment and sustainable work life?

OTHER OUTCOMES:
Background data | descriptive data at baseline= one measurement
  Age, gender, profession, number of years working in the profession, public/private dental clinic, working hours,
Semi-structured individual interview study with managers, sub-study 2 | Baseline=one interview
  Open questions following the interview guide described above under the study description section

CONTACTS AND LOCATIONS:
Overall Officials: Anneli Peolsson, Professor, Principal Investigator — Occupational and Environmental Medicine Center, Linköping University, Linköping, Sweden
Locations (1):
- Occupational and Environmental Medicine Centre, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Coded data will be available open reasonable request and after ethical permission (because of health data).
Supporting Information: Study Protocol
Time Frame: After data is collected and published.
Access Criteria: Coded data will be available open reasonable request and after ethical permission.